CLINICAL TRIAL: NCT05832398
Title: Precision Chemotherapy Based on Organoid for Colorectal CancerPatient-Derived Tumor Organoid Drug Sensitivity for Colorectal Cancer: A Prospective, Multicentre，Randomized, Controlled Trial
Brief Title: Precision Chemotherapy Based on Organoid Drug Sensitivity for Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-471
Record Dates: First submitted 2023-02-06; First posted 2023-04-27 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: Organoid; Drug Test
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Oxaliplatin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organoid guided chemotherapy (Experimental): Patients will receive sensitive chemotherapy in organoid drug test once every two weeks for 6 cycles as adjuvant chemotherapy
  Interventions: Drug: FOLFOX , FOLFIRI or FOLFOXIRI regimens
- FOLFOX regimen (Active Comparator): Patients will receive FOLFOX regimen once every two weeks for 6 cycles as adjuvant chemotherapy
  Interventions: Drug: FOLFOX or CapeOX regimens

INTERVENTIONS:
Drug: FOLFOX , FOLFIRI or FOLFOXIRI regimens — FOLFOX (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 400mg/m2 infusion, and 2400mg/m2 as a 46-hour continuous infusion on day 1) for 6 cycle FOLFIRI (irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 400mg/m2 infusion, and 2400mg/m2 as a 46-hour continuous infusion on day 1) for 6 cycle FOLFOXIRI (irinotecan 150mg/m2, and folinic acid 400mg/m2, oxaliplatin 85 mg/m2, 5-fluorouracil 3200 mg/m2 48-h continuous infusion) for 6 cycle
  Other Names: oxaliplatin, irinotecan, 5-fluorouracil
  Arms: Organoid guided chemotherapy
Drug: FOLFOX or CapeOX regimens — FOLFOX (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 400mg/m2 infusion, and 2400mg/m2 as a 46-hour continuous infusion on day 1) for 6 cycle CaoeOX (Oxaliplatin 130 mg/m2 intravenous infusion on day 1,Capecitabine 1000 mg/m2 twice daily PO for 14 days)
  Other Names: oxaliplatin, 5-fluorouracil
  Arms: FOLFOX regimen

SUMMARY:
The purpose of this study is to investigate whether chemotherapy guided by patient-derived tumor organoid drug test can improve the outcomes of stage IV colorectal cancer.

DETAILED DESCRIPTION:
Fluorouracil-based chemotherapy is the standard treatment for stage IV colorectal cancer patients. However, the effects of chemotherapy remains limited. Patient-derived tumor organoids are increasingly used as tools for drug test and predicting drug response in the clinic, and have been showed to faithfully predict clinical outcomes of patients with CRC. A prospective clinical trial is needed to validate whether the in vitro sensitivity to chemotherapy regimens in organoids drug test is associated with a longer PFS in stage IV colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Histological confirmed colorectal cancer
* Stage IV
* American Society of Anesthesiologists (ASA) score I~III
* No contraindication for chemotherapy
* No evidence of other malignant tumor

Exclusion Criteria:

* Refusing chemotherapy
* Pregnant or breast-feeding women
* Severe organ damage after chemotherapy, surgery or unable to continue to systemic chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Progression-free survival | up to 1 years
  the time from randomization to relapse or death, whichever occurred first

SECONDARY OUTCOMES:
Overall survival | up to 5 years
  the time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yan, M.D., Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No